CLINICAL TRIAL: NCT06884917
Title: The Effect of Sleep Hygiene Education Based on the Comfort Theory of Kolcaba Given to Menopausal Women on Comfort Behaviors and Sleep Quality
Brief Title: Effect of Sleep Hygiene Education on Comfort and Sleep Quality in Menopausal Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 211002081
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-02

CONDITIONS: Women in the Menopausal Period
Keywords: Comfort; Menopause; Sleep Hygiene; Sleep Quality
MeSH Terms: conditions — Sleep Hygiene; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Hygiene Training (Experimental): Women who will participate in the Sleep Hygiene Education based on Comfort Theory (intervention group) will have face-to-face meetings in the meeting rooms of Zeynep Kâmil Women's and Children's Diseases Training and Research Hospital. The date and time of the meetings will be scheduled according to the women's availability and they will be contacted a day before the scheduled training day as a reminder. If the women do not attend the appointment, a new appointment will be scheduled for another day. A total of three meetings will be held with each woman, each lasting 60 minutes. Looking at the intervals between the meetings; the first and second sessions will have a two-week gap, and there will be an eight-week gap between the second and third sessions. The first measurement will be taken before the first meeting, and the final measurement will be conducted after the third meeting. After the second meeting, a brochure on sleep hygiene will be provided.
  Interventions: Other: Sleep Hygiene Training
- Observation (No Intervention): The control group will be given the first measurement before the first interview of the intervention group and the last measurement after the third interview of the intervention group. The control group will be given a brochure on sleep hygiene after the third interview.

INTERVENTIONS:
Other: Sleep Hygiene Training — Written consent will be obtained from the women, and a Personal Information Form will be applied. The General Comfort Scale (GCS) will be applied to the women. The Pittsburgh Sleep Quality Index (PSQI) will be applied to the women. Each level will include the physical, socio-cultural, psycho-spiritual, and environmental dimensions where the requirements to ensure comfort arise.
  Arms: Sleep Hygiene Training

SUMMARY:
The decrease in estrogen levels in the body during menopause can lead to sleep disturbances by disrupting serotonin metabolism, which plays an important role in regular sleep. Considering the increase in life expectancy, the duration of time women will spend in menopause is also increasing, making the understanding of menopause physiology and potential management strategies highly important for women's health.

One of the most important factors in managing insomnia is sleep hygiene. Sleep hygiene is defined as the principles and practices that improve sleep quality. Additionally, during menopause, using the comfort theory to recognize unmet comfort needs, collecting data on these needs, providing interventions, and ensuring the individual's comfort at the highest level are responsibilities of the nurse. To achieve this, the nurse needs to determine the individual's comfort level before providing care, then assess their physical, psychosocial, sociocultural, and environmental comfort needs as a whole.

This research is designed as a randomized pre-test post-test control group study to evaluate the impact of Kolcaba's comfort theory-based sleep hygiene education on comfort behaviors and sleep quality in menopausal women. The research will be conducted between July and December 2024 at Zeynep Kâmil Women's and Children's Diseases Training and Research Hospital, Gynecology Outpatient Clinic, in Istanbul. The study population will consist of menopausal women who visit the Gynecology Outpatient Clinic. The sample will include premenopausal women who meet the inclusion criteria for the study. The sample size in the study was planned to be 60 (intervention group = 30, control group = 30), calculated using the G Power version 3.1 program with α = 0.05, 1-β = 0.95, and effect size = 1.00, considering the possibility of sample loss.

Data will be collected using the "Personal Information Form (Appendix-1)", "General Comfort Scale (Appendix-2)", and "Pittsburgh Sleep Quality Index (Appendix-3)". The data will be analyzed using SPSS 22.0 software.

A total of three sessions will be conducted with each woman, with each session lasting 60 minutes. The intervals between sessions will be arranged as two weeks between the first and second sessions, and eight weeks between the second and third sessions. The first measurement will be taken before the first session, and the final measurement will be taken after the third session.

DETAILED DESCRIPTION:
1. MENOPAUSE PERIOD The life stage following women's sexual maturity is called the "Climacteric Period." The climacteric period is a phase during which physical, psychological, and social changes occur, and certain health problems may arise. The most significant change of this period is menopause. The term menopause, which originates from the Greek words "men" (month) and "pausis" (cessation), is defined as the permanent cessation of menstrual bleeding, diagnosed after 12 months of amenorrhea, and not explainable by pathological or hormonal causes. The basic mechanism is related to a decrease in estrogen levels and an increase in follicle-stimulating hormone (FSH) levels. Menopause is an important life phase marking the end of women's natural reproductive cycle, with the average age of menopause being 51. The period 2-6 years before menopause is called the premenopausal period, and 6-8 years after menopause is called the postmenopausal period. The perimenopausal period, which is the transition period to menopause, begins with menstrual irregularities and includes the early postmenopausal period following the last menstrual period.

   During menopause, women experience numerous complaints such as hot flashes, night sweats, weight gain, vaginal dryness, thinning of the skin, sleep disturbances, psychological changes, and osteoporosis. These symptoms cause physiological, mental, social, and sexual changes in women. These complaints, which begin in the premenopausal period, arise due to fluctuations in sex hormone levels during the follicular and luteal phases of the menstrual cycle, whereas in the postmenopausal period, they can appear due to the absence of estrogen.

   With the increase in life expectancy at birth, the duration that women spend in the menopausal period is increasing, making it crucial to understand the physiology of menopause and potential management strategies for women's health. Moreover, menopause occurs during a critical period in women's lives, coinciding with various social transitions, such as children leaving home, and women experiencing "Empty Nest Syndrome," where they feel more isolated with increasing psychosomatic symptoms. In other words, the menopausal symptoms experienced during and after the transition to menopause vary from woman to woman. While some women do not report symptoms, for others, these symptoms can be severe and negatively impact their daily activities and quality of life. The presence and severity of these symptoms can vary greatly, lasting from months to years.

   1.1. Changes Seen During Menopause After menopause, numerous physiological, psychological, and behavioral changes occur in women. Approximately 85% of women experience symptoms during menopause. These symptoms generally include vasomotor symptoms, sleep disturbances, emotional changes, hair and skin changes, urogenital changes, sexual changes, metabolic syndrome, cardiovascular changes, gastrointestinal changes, and musculoskeletal system changes.

   The most common menopausal symptoms due to estrogen deficiency are vasomotor changes, which include hot flashes, night sweats, and hot flushes. Hot flashes are often accompanied by sweating, anxiety, chills, and palpitations. These symptoms can affect a woman's daily life. The severity of symptoms tends to decrease as time passes after menopause. Hot flashes can be triggered by crowded, hot environments, alcohol, hot beverages, spicy foods, emotional stress, caffeine, certain medications, and smoking.

   Hormonal changes during menopause are known to cause various psychological changes, affecting mood and behavior. Psychological symptoms associated with menopause include feelings of depression, irritability, worthlessness, difficulty making decisions, anxiety, forgetfulness, difficulty concentrating, feelings of inadequacy, fatigue, decreased sexual desire, frequent crying, anxiety, being easily affected by daily events, increased appetite, general lack of interest, sleep disturbances, and waking up early in the morning, as well as social withdrawal.

   Urogenital organ atrophy develops due to estrogen deficiency. As a result, vaginal dryness occurs because of reduced vaginal blood circulation. The atrophic vagina loses its elasticity, becomes pale, pubic hair decreases, and the vagina narrows and becomes fragile. Vaginal discharge decreases, and dyspareunia may occur due to dryness. During this period, the vaginal pH increases, leading to increased susceptibility to infections. Urinary complaints also increase, and conditions such as vaginitis, urovaginal prolapse, rectocele, and cystocele may be observed.

   Hormonal changes affect metabolism, leading to an increase in total body fat percentage, especially around the abdominal area, which increases the risk of obesity. Changes in fat metabolism lead to an increased risk of hypertension and heart diseases. Estrogen deficiency causes changes in bone metabolism, reducing calcium and phosphorus absorption, which can lead to osteoporosis.

   One of the most common complaints during menopause is sleep problems, which become more prevalent and often troublesome during both premenopausal and postmenopausal periods. Due to the decrease in estrogen levels during menopause, the serotonin metabolism, which plays an essential role in regular sleep, is disrupted. This results in a reduction in total sleep duration and an increase in sleep onset latency, which can lead to sleep disturbances. Endogenous melatonin secretion decreases with age and varies by gender. In menopausal women, melatonin levels decrease significantly, affecting sleep patterns. Progesterone has a general protective effect on sleep apnea in women of reproductive age. It activates benzodiazepine receptors and gamma-aminobutyric acid receptors, which induce sleep and have anxiolytic effects. The decline in progesterone levels during menopause is associated with sleep disorders.

   Sleep disturbances are seen in 40-60% of perimenopausal and postmenopausal women, and they often persist in later stages. Studies have shown that postmenopausal women have more difficulty falling asleep and experience sleep apnea more often than perimenopausal women. Another study found that although total sleep duration was similar in premenopausal and postmenopausal women, it was shorter than in younger women. Sleep efficiency was found to be 93.4% in young women, 84.3% in perimenopausal women, and 80.2% in postmenopausal women. Perimenopausal and postmenopausal women tend to wake up more often during the night, with insomnia being more frequent, especially in the postmenopausal period.

   The most common sleep disorders among menopausal women are insomnia, sleep apnea, and restless leg syndrome. These sleep disorders are more common during the menopausal period and can lead to physical and psychological conditions such as cardiovascular diseases, diabetes, depression, anxiety, and the excessive use/abuse of hypnotic medications. Therefore, understanding sleep physiology and managing sleep disorders is crucial. Menopausal women should be carefully evaluated by a multidisciplinary team, addressing both psychological and somatic symptoms.
2. SLEEP AND SLEEP PHYSIOLOGY Sleep is a dynamic process that serves as both a resting and preparing phase for the body's physiological and psychological regulation. This dynamic process, which is expected to occur daily, plays a key role in both physical and mental health. In the natural sleep cycle, there are two specific areas controlled by the brainstem: the Reticular Activating System (RAS) in the cerebral cortex and the Bulbar Synchronizing System (BSR) in the medulla. These two systems work in synchrony. The RAS is responsible for cortical activities associated with wakefulness, as well as reflex and voluntary movements. During sleep, it can detect stimuli such as pain, noise, or pressure from the periphery and the cerebral cortex, causing the individual to wake up.

   As stimuli decrease, the activation of the RAS also diminishes. Serotonin plays a significant role in regulating sleep. It is secreted from the Rafe nuclei within the RAS. If this nucleus is damaged or serotonin synthesis is inhibited, sleep duration decreases. During the sleep process, in addition to serotonin release, body temperature and serum cortisol levels decrease, while melatonin secretion increases. As norepinephrine is inhibited in the subcortical region of the central nervous system, the body prepares for sleep. With the increase in serotonin levels, sleep deepens, and as sleep deepens, inhibition of the adrenergic system increases. Increased activity in the BSR area initiates sleep. In other words, the transition from wakefulness to sleep is achieved by inhibiting RAS and increasing BSR activation.

   2.1. Sleep Stages Sleep consists of two phases: NREM (Non-Rapid Eye Movement) sleep, also known as slow-wave sleep, and REM (Rapid Eye Movement) sleep. These phases alternate throughout the sleep process in cycles.

   NREM (Non-Rapid Eye Movement) Stage: This stage constitutes approximately 75% of sleep. During this stage, brain waves slow down, and rapid eye movements are absent. Each cycle lasts about 90 minutes, with 4-6 cycles occurring throughout the night. NREM begins with the onset of sleep and represents deep, restorative sleep, characterized by a decrease in physical and psychological activity, and the absence of rapid eye movements. During NREM sleep, heart rate and respiration slow by 20-30%, blood pressure drops, muscles relax, heat loss increases, metabolic rate slows by 10-30%, and body temperature decreases.

   REM (Rapid Eye Movement) Stage: This phase constitutes about 15-25% of sleep and is considered the active phase of sleep, characterized by rapid eye movements. REM cycles last 5-30 minutes and repeat every 80-100 minutes. In this phase, autonomic nervous system activity increases, leading to irregularities in respiration, cardiac rate, and blood pressure. REM is involved in the genetic programming of learning and is considered the period for mental relaxation.

   2.2. Functions of Sleep and Factors Affecting Sleep Sleep is one of the most crucial physiological processes for maintaining and sustaining physical and mental well-being. Quality sleep directly affects daily life, emotional and social well-being, and overall quality of life. The potential functions of sleep include body rest and preparation for the next day, energy storage, growth, protection, cell rejuvenation, body renewal, revitalization, consolidation of learned information, prevention of corneal anoxia, maintenance of neuronal integrity, and adaptation to the environment, especially in some animals.

   A study in Turkey revealed that 75% of the population sleeps 7-8 hours per day, while 10% sleep only 6 hours. There are varying opinions regarding the function of sleep. Some suggest that sleep is a state where all behavioral and physiological responses of the organism slow down, the sensory gates close, and the organism is protected. Meanwhile, others suggest that sleep is an active process in which the brain works actively to repair and restore itself, process learned information, and prepare the brain cortex for wakefulness.

   Various factors can affect sleep quality, including age, gender, health conditions, medication, alcohol and stimulant use, lifestyle, exercise, fatigue, anxiety, stress, diet, occupation, economic status, working conditions, and established habits. Impaired sleep quality can lead to metabolic issues such as insulin resistance and increased diabetes risk, disturbances in growth.
3. SLEEP HYGIENE In addition to sleep disorders and medical issues, daily behaviors, routines, and environmental exposures related to noise, temperature, sleep surface, and light exposure also play an important role in sleep. Individuals may use sleeping pills or alcohol to induce sleep. Sedative agents such as benzodiazepines, antihistamines, alcohol, and barbiturates can help with sedation, but they are also associated with negative outcomes, including physical and mental dependency, non-physiological sleep, daytime sedation, behavioral side effects, and increased risks of falls and mortality, especially during menopause and in the elderly population. In the long term, the best treatment for improving sleep involves behavior changes that include routines promoting healthy sleep. Sleep hygiene refers to behavioral and lifestyle interventions that positively affect sleep duration and sleep quality throughout the day. Sleep hygiene is addressed under behavioral therapies.

   The necessary daily practices, habits, and environmental adjustments to improve sleep quality at night are covered under sleep hygiene. Sleep hygiene education is commonly used as a coping strategy for sleep disorders. Sleep hygiene adjustments are an effective and inexpensive approach in the management of sleep disorders, without side effects. Sleep environment, regulating sleep time, daily activities, and food intake, and improving mental control behaviors are sub-dimensions of sleep hygiene education.

   3.1. Regulation of the Sleep Environment The main environmental factors that are effective in falling asleep and maintaining sleep are noise, room temperature, presence of stimuli, and light conditions. Therefore, optimizing the bedroom environment can enhance sleep quality. Thermal environment is one of the important factors affecting sleep. Extremely hot or cold rooms make it difficult to fall asleep, increase wakefulness, and reduce REM sleep and slow-wave sleep. The effect of the thermal environment on sleep cycles is closely related to thermoregulation mechanisms that influence sleep-regulating mechanisms. A cold environment affects cardiac autonomic responses and thus influences sleep.

   When individuals are exposed to light before sleep, a signal is sent to the brain through a reduction in melatonin secretion. Even low levels of light reflected from phones or e-readers can delay sleep and make it harder to wake up the next morning. Reducing both ambient light and light from electronic devices makes it easier to fall asleep and improves sleep quality. Approaches to reduce light exposure include avoiding screens, dark rooms, blue-light blocking glasses, and sleep masks.

   Because the brain processes auditory stimuli both in wakefulness and sleep, sleep quality can be affected by auditory pollution. When noise levels range from 40 to 55 dB, individuals typically try to adjust their environment to maintain adequate sleep quality. However, when noise levels exceed 55 dB, sleep problems become more frequent. White noise machines or earplugs can be used to block noise. Additionally, avoiding using the bed for work, watching TV, and other non-sleep activities can also be helpful.

   Pillow comfort can also affect sleep quality, as a well-designed pillow allows more surface contact with the neck, enabling more even pressure distribution on the cervical (neck) muscles. There is no recommended sleep surface, sleep position, or pillow. Individuals are advised to use a mattress, pillow, and bedding that are most comfortable and find the sleep position that works best for them. However, individuals with untreated sleep apnea are advised to avoid sleeping on their backs. Mattress comfort can also affect sleep quality by facilitating position changes throughout the night, helping to prevent muscle stiffness. Studies in adults with chronic pain suggest that a moderately firm mattress may be beneficial for optimizing sleep, regardless of age.

   3.2. Regulation of Sleep Timing Adequate sleep is essential for health, and individuals are recommended to sleep for an average of 7-8 hours per night. Sleeping less than seven hours is associated with negative health outcomes, including weakened immune system, performance impairment, increased errors, and a higher risk of accidents. Going to bed and waking up at the same time every day improves circadian rhythm synchronization and enhances sleep quality. In cases where the time spent sitting up at night is extended, it becomes more difficult to fall asleep, sleep duration decreases, and insufficient sleep occurs. In menopausal women, irregular sleep schedules and late bedtimes are more likely to result in insomnia.

   Sleeping and waking up at the same time every day, including weekends and during travel, is one of the most important elements of sleep hygiene. A regular sleep schedule helps maintain the body's circadian rhythm, reduces daytime sleepiness, and makes it easier to fall asleep and wake up. Additionally, aligning with the circadian rhythm helps regulate mental health, the endocrine system, and the reproductive system. Studies suggest that when individuals fail to align with the circadian rhythm, negative health outcomes such as metabolic disorders, cardiovascular diseases, immune system disorders, cancer, and mental health deterioration become more frequent.

   Meta-analysis studies have shown that a single sleep period of 7-8 hours in darkness with a regular schedule is optimal. However, research also shows that short sleep periods, called naps, can provide important health benefits, such as relaxation, reduced fatigue, improved mood, and increased alertness. Afternoon naps lasting 20-30 minutes are typically the most suitable. Longer naps, if the individual enters deep sleep, can lead to grogginess or disorientation upon waking. In menopause and old age, excessive napping has been associated with negative outcomes. If an individual has sleep problems, short nap periods should not be recommended, as they can lead to delays in the desired bedtime and more difficulty falling asleep.

   3.3. Regulation of Daily Activities Regular exercise positively affects sleep health. Exercise raises body temperature. Two to four hours after exercise, body temperature drops, which helps to fall asleep and maintain sleep. At the same time, exercise is perceived as a physical stressor by the body, and the body responds by increasing deep sleep. Regular exercise activates the endocrine system and regulates hormonal fluctuations in women. The National Sleep Foundation encourages exercise at any time of day, without any restrictions. While the exact mechanism through which physical activity improves sleep is unclear, studies have shown that moderate aerobic exercise is beneficial, increasing deep sleep and sleep duration. Exercise has also been shown to reduce pre-sleep anxiety and improve sleep in individuals with chronic primary insomnia.

   3.4. Regulation of Food Intake Obese individuals (with a body mass index greater than 30 kg/m2) report subjective sleep problems twice as often as non-obese individuals. Being obese or overweight is associated with a reduction in sleep duration compared to non-obese individuals. Major factors contributing to obesity include environment, eating behavior, physical inactivity, psychosocial conditions, and genetics. Additionally, overweight or obesity rates are higher in menopausal women compared to men. Based on these factors, losing weight or maintaining an optimal body weight may help reduce sleep problems. For example, weight loss has been shown to significantly improve sleep disorders such as sleep apnea, increase sleep quality, and reduce daytime sleepiness.

   Inadequate sleep and excessive calorie intake can cause hormonal imbalances. One of these imbalances is a decrease in melatonin levels, which causes changes in metabolic circadian rhythms, leading to weight gain and metabolic syndrome. There are also changes in the effects of leptin and insulin hormones. Obese individuals develop resistance to both of these hormones. These hormones reduce food intake and increase energy metabolism. Ghrelin, secreted by the stomach, stimulates appetite and is also affected by sleep disorders. Changes in these levels in individuals with insomnia lead to increased food intake and contribute to obesity.

   Milk and dairy products are rich in specific casein hydrolysate, tryptophan, and magnesium, which are beneficial in reducing sleep disorders. Studies have found that drinking milk or eating cheese makes it easier to fall asleep. Research shows that eating late at night is associated with later bedtimes, shorter sleep duration, and weight gain. It is recommended that individuals avoid eating within two hours of bedtime, if possible. Avoiding large, mixed meals and unhealthy foods before sleep can help improve sleep quality and prevent weight gain.

   Caffeine is a stimulant with effects that can diffuse throughout the body, pass the blood-brain and placental barriers, and disrupt sleep. Caffeine is an antagonist of adenosine receptors, and for this reason, it is a cause of sleep disturbances. Caffeine reduces sleep onset time, total sleep time, and sleep quality, leading to insomnia. Menopausal and elderly individuals may be more sensitive to caffeine, and genes associated with adenosine neurotransmission may influence individual sensitivity to caffeine-induced sleep deprivation. Due to genetic variation, the half-life of caffeine is 6-7 hours. As a result, avoiding caffeine after midday can help increase the likelihood of falling asleep when desired.

   Alcohol is theoretically a sedative that helps individuals fall asleep. However, it can disrupt sleep patterns and often causes waking in the second half of the night. While alcohol reduces deep sleep and REM sleep during the first hours of sleep, it increases REM sleep and nighttime awakenings in the later hours. Individuals who use alcohol to help them sleep are at risk for substance dependence issues and liver damage. Additionally, there may be a fine line between passing out and falling asleep. Chronic alcoholism leads to temporary and permanent changes in brain systems that regulate sleep. Alcohol affects adenosine release, causing sleep disturbances. Alcoholics often complain of deep sleep deprivation, daytime sleepiness, and altered sleep patterns.

   Nicotine, contained in cigarettes, has a stimulating effect. Due to this effect, individuals may have difficulty falling asleep. A drop in nicotine levels several hours after falling asleep can disrupt sleep, reduce restorative deep sleep, and shorten sleep duration. Two sleep disorders commonly associated with smoking are insomnia and sleep apnea. Studies have found that smokers experience sleep problems 1.45 times more frequently than non-smokers. Smokers are more likely to experience a drop in oxygen saturation, increased airway resistance, and inflammation, all of which contribute to the development of sleep apnea.

   3.5. Regulation of Mental Control Suppression of the hypothalamic-pituitary-adrenal axis is a factor that facilitates falling asleep. Insomnia is often characterized by deep thinking associated with serious and undesirable activation of the autonomic nervous system. Stress activates the hypothalamo-pituitary-adrenal axis, causing sleep disturbances. Studies have shown that insomnia symptoms are 1.7 times more frequent in chronic moderate to severe stress conditions, and another study found that stress reduces sleep duration. High levels of stress lead to an increase in depressive symptoms, increased severity of weakness, and a reduction in total sleep time. Yoga is known to reduce perceived stress and improve sleep quality. In a study by Jespersen and colleagues (2022), relaxation techniques combined with music were found to improve total sleep time and sleep efficiency. Deep breathing and relaxation exercises, done for relaxation, send signals to the nervous system, slowing neuronal activity and heart rate, and thus advancing sleep.
4. Kolcaba's Comfort Theory The concept of "comfort" is derived from the Latin word "confortare," meaning "to strengthen." In the Oxford English Dictionary, it is defined as "the state of physical and material well-being by meeting bodily needs and relief from discomfort and pain," "relief from mental distress or anguish and receiving support," "comforting, soothing," and "strengthening, encouraging, and helping." According to Kolcaba, comfort is "an expected outcome with a complex structure in the context of physical, psychospiritual, social, and environmental integrity, helping to meet the individual's needs, providing peace, and overcoming problems." According to the holistic approach, Kolcaba defines the concept of comfort as "the experience of meeting basic human needs to achieve relief, peace, and the ability to overcome problems in the present moment."

   The Comfort Theory was first introduced as a nursing theory in 1990 by Katharina Kolcaba. Kolcaba continued her studies on the concept of comfort and the provision of patient comfort for approximately 15 years and, in 1988, developed the taxonomic structure of comfort, consisting of three levels and four dimensions. The basic assumptions of the Comfort Theory are as follows:
   * Individuals respond to complex stimuli holistically.
   * Comfort is a desired outcome specific to nursing.
   * Individuals must meet basic comfort needs themselves, or these needs must be met by others.
   * Traditional integrity has a rule-based and descriptive structure rooted in a patient-centered value system.

   After completing the conceptual studies on comfort, Kolcaba began developing the General Comfort Questionnaire (GCQ), a 48-item Likert-type scale, to measure the expected comfort outcome in patients and published the results in 1992.

   4.1. Concepts of Comfort Theory As a result of her work on comfort and patient comfort, Kolcaba developed the taxonomic structure of the Comfort Theory, which consists of three levels and four dimensions. The Comfort Theory includes three levels: Relief, Ease, and Transcendence.

   Relief: This refers to the feeling of relief from a situation that disrupts comfort. It is described as the state of the individual feeling relieved as a result of meeting their needs. Relief occurs when a specific need is met and is necessary for returning to previous functions or peaceful death. Derived from nursing theories, relief is a feeling experienced by patients whose needs are met according to Orlando's theory, and is described in Henderson's theory as the feeling that occurs when any of the 14 basic needs of the patient are met.

   Ease: This is the state of being comfortable. It is defined as the state of being calm, relaxed, or at peace. The patient's ease is expressed by their satisfaction and the indication that they are content. It is influenced by the individual's physical and emotional experiences, as well as environmental factors.

   Transcendence: This refers to personal growth and the feeling of renewal. It is defined as the situation where the individual overcomes problems and enhances their ordinary powers. An individual whose comfort needs are fully met reaches the level of transcendence, which is the ability to overcome problems. All three comfort levels positively influence the performance of the patient and are theoretically empowering components.

   The dimensions of the Comfort Theory include the physical, socio-cultural, psychospiritual, and environmental environments where comfort-related needs arise.

   Physical Comfort: This relates to bodily perceptions. It includes physiological factors such as rest and relaxation, responses to illness, nutrition and homeodynamics, and the continuity of bowel functions that affect the individual's physical condition. Pain is considered one of the biggest factors that reduce physical comfort. Whether or not it creates a stimulus, physical comfort is formed by the individual's responses to illnesses. In this sense, the necessary physiological indicators for physical comfort include fluid-electrolyte balance, regular and balanced blood chemistry, adequate oxygen saturation, and metabolic reactions. Any deviation from the normal in one of these physiological indicators may affect comfort.

   Psychospiritual Comfort: This involves cognitive, spiritual, and emotional components. It encompasses elements that give meaning to the individual's life, such as self-respect, self-concept, sexuality, and awareness of self.

   Environmental Comfort: This encompasses external factors, situations, and their effects on the individual. Concepts related to the individual's external environment, such as lighting, noise, room color, room temperature, a safe environment, and the view from the window, are included in environmental comfort.

   Socio-Cultural Comfort: This includes providing information and counseling, offering care sensitive to the individual's/family's traditions and habits, religious beliefs, using financial support systems, facilitating interpersonal communication, discharge planning, discharge education, and providing home care. These are the factors that form socio-cultural comfort.

   When the taxonomic structure of Comfort Theory is examined, each component is interconnected. For example, physical comfort relates to bodily perceptions. Therefore, when the individual's needs for various stimuli are met, they will be relieved of the discomfort caused by those responses and achieve the desired comfort level.
5. Sleep Hygiene Education Based on Comfort Theory Nursing care has an important quality in orienting an individual who experiences physical and psychosocial problems, preventing these problems, treating them, and ensuring comfort. Nurses are also responsible for providing comfort to individuals. The primary aim of nursing interventions is to increase the comfort of individuals. An individual who cannot be comforted feels a sense of deficiency. On the other hand, individuals who are comfortable and free of discomfort recover more quickly, cope better with illness-related stress, and rehabilitate more effectively.

There is a direct relationship between meeting an individual's needs and ensuring their comfort. By utilizing Comfort Theory, recognizing unmet comfort needs of the individual, collecting data on these needs, intervening, and maintaining the highest level of comfort are the nurse's responsibilities. To achieve this, the nurse should first determine the individual's pre-care comfort level, then assess the individual's physical, psychospiritual, sociocultural, and environmental comfort needs by considering them as a whole. Afterward, the nurse should implement nursing interventions to enhance comfort for unmet needs, evaluate the results, and, if necessary, make new plans. Providing nursing care to ensure comfort, along with evaluating the expected comfort outcome, has been shown in studies to impact the quality of care, individual satisfaction, and quality of life. Reducing uncertainty and increasing comfort levels requires identifying individuals' care needs and implementing nursing interventions based on these needs. The individual lives in a bio-psycho-social-environmental-spiritual integrity. One of the most fundamental concepts in nursing care is the holistic approach. This approach requires understanding that the bio-psycho-social-environmental-spiritual dimensions interact with each other, and when one dimension is not properly addressed, the individual's health condition may deteriorate. During menopause, sleep hygiene education should be given to the individual in a holistic way. The components of holistic care in sleep hygiene education during menopause are as follows:

* Physical care
* Psychospiritual care
* Sociocultural care
* Environmental care.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agree to participate in the study, Are literate, Are open to communication and cooperation, Score 5 or higher on the Pittsburgh Sleep Quality Index (PSQI), Have a Body Mass Index (BMI) lower than 30 kg/m², Have one or more of the following symptoms: vasomotor symptoms such as hot flashes and night sweats, menstrual irregularities, vaginal dryness, urinary incontinence, or sleep disturbances, Are in the premenopausal period and have consulted the gynecology outpatient clinic.

Exclusion Criteria:

* Diagnosed with a sleep disorder, Have a chronic illness, Are undergoing hormone replacement therapy, Use sleep-related medications such as melatonin, benzodiazepines, antihistamines, and barbiturates, Use alcohol or cigarettes.

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Premenopausal women who present to the gynaecology outpatient clinic with one or more of the following symptoms: vasomotor symptoms such as hot flushes, night sweats, menstrual irregularities, urogenital symptoms such as vaginal dryness, urinary incontinence, sleep disorders such as disturbed sleep patterns.
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
General Comfort Scale (GCS) | Through study completion, an average of 6 months
  The General Comfort Scale was developed by Kolcaba in 1992. It is used to assess the increase in comfort expected from nursing interventions that promote comfort by identifying individual needs. The scale is a four-point Likert type and contains a total of 48 items. The scale consists of both positive and negative items, with the response patterns mixed. In this regard, a high score (4) on positive items indicates high comfort, and a low score (1) indicates low comfort. In the evaluation of the scale, the negative scores are reverse-coded and summed with the positive items. The highest total score that can be obtained from the scale is 192, and the lowest total score is 48. The Turkish validity and reliability of the scale were conducted by Kuğuoğlu and Karabacak in 2004. In the internal consistency analysis of the scale, Kuğuoğlu and Karabacak (2008) found the Cronbach's Alpha coefficient to be 0.85 and reported that the scale has high reliability.
Pittsburgh Sleep Quality Index (PSQI) | Through study completion, an average of 6 months
  The PSQI was developed by Buysse and colleagues in 1989. The validity and reliability study of the PSQI was conducted by Ağargün and colleagues in 1996, and the Cronbach Alpha value was calculated to be 0.79. The PSQI is a self-report scale that evaluates sleep quality and disturbances over a one-month period. The scale consists of seven subcomponents: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medications, and daytime dysfunction. It includes a total of 24 questions, with the first 19 questions answered by the individual, and the last five questions answered by the individual's bed partner or roommate. Each item in the scale is scored between 0 and 3, and the total score ranges from 0 to 21. Higher scores indicate poor sleep quality and a higher level of sleep disturbance. A total score of over five indicates clinically poor sleep quality.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Sağlık Bilimleri Ünversitesi, Istanbul, Türkiye
  - Sağlık Bilimleri Ünversitesi, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided